CLINICAL TRIAL: NCT00516204
Title: Diabetic Under 70 (Diabetics Below 70)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CAT-CRE-2007/3; NIS-CAT-DUM-2007/3
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes; Hyperlipidemia; Atherosclerosis
Keywords: Hyperlipidemia; Diabetics; NIS; Diabetics with hyperlipidemia and atherosclerosis (coronary heart disease, carotid stenosis, PAVK, etc.)
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias; Atherosclerosis; Coronary Disease; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (4):
- Patients at very high risk
- Patients at high risk
- Patients at medium risk
- Patients at low risk

SUMMARY:
A screening project of diabetics with a very high cardiovascular risk (e.g. diabetes plus coronary heart disease) who already receive cholesterol-lowering therapy. Lipid profile and rate of patients who are treated to target (which is <70mg/dl for such patients with very high risk) are screened. The doctors therapy decisions after the screening will be documented and 8-10 weeks later the lipid profile of each patient will be evaluated again. Our aim is to evaluate dosing habits, to evaluate how many patients are treated to their LDL-C target and to underline the importance of treating patients to their cholesterol targets.

ELIGIBILITY:
Inclusion Criteria:

* Diabetics with hyperlipidemia and atherosclerosis (coronary heart disease, carotid stenosis, PAVK, etc.) who already receive cholesterol-lowering therapy

Exclusion Criteria:

* Diabetics w/o CVD; diabetics who do not receive cholesterol-lowering therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female secondary prevention patients with: coronary disease with event: acute coronary syndrome, status post MI, PTCA, CABG, angiographically verified), PAVK (min. IIb or S.p. revascularization), stroke/TIA, carotis-plaque (asymptomatic min. 70% or S.p. revascularization), Diabetes Mellitus (type I, II)
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2007-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cholesterol levels | After 4 weeks
  Cholesterol levels from high risk patients after 4 weeks of cholesterol-lowering drug therapy under target values

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, MD, Study Chair — Chairs of the Austrian Diabetes Society
Locations (1):
- Research Site, Vienna, Austria